CLINICAL TRIAL: NCT06767696
Title: The Effect of Neck Hyperextension on Endotracheal Tube Cuff Pressure in Children
Brief Title: Effect of Neck Hyperextension on Endotracheal Tube Cuff Pressure in Children
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ERBİL TÜRKSAL, Medical Doctor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BÇEK/163
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Endotracheal Cuff; Adenoidectomy Surgery; Tonsillectomy with or Without Adenoidectomy; Position Differences

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paediatric patients with adenoidectomy and/or tonsillectomy: Patients aged 2-18 years undergoing adenoidectomy, tonsillectomy or adenotonsillectomy surgery during the study period
  Interventions: Other: Cuff pressure measurement

INTERVENTIONS:
Other: Cuff pressure measurement — Intubation tube cuff pressure in cmH2O at 3 different time periods with a cuff manometer (VBM Medizintechnik, GmbH, Germany)
  Time periods:
  Cuff pressure value measured in neutral position after intubation (cmH2O) - T0 Cuff pressure measurement value after hyperextension (cmH2O) - T1 Cuff pressure measurement value in neutral position after surgical procedure (cmH2O) - T2

SUMMARY:
Introduction: Patients undergoing surgery under general anaesthesia are frequently intubated with an endotracheal tube (ETT). The safety margin of ETT cuff pressure is between 20-30 cmH2O. Inadequately inflated cuff (<20 cmH2O) may cause secretions in the mouth, foreign bodies, bleeding due to surgery to escape into the trachea and/or air leakage. As a result of air leakage, the effect of mechanical ventilation decreases, end-tidal CO2 measurement cannot be performed accurately, and inhalation anaesthetics leak into the operating room. An overinflated cuff (>30 cmH2O) may affect tracheal mucosa blood flow. This may result in tracheal stenosis, tracheoesophageal fistula or tracheal rupture. There may be significant changes in cuff pressure during endotracheal intubation because cuff pressure can be affected by changes in head and neck position. Due to all these situations, controlling ETT cuff pressure is very important for patient health and safety.

For ETT cuff pressure control; manual palpation of the pilot balloon, listening for the disappearance of an audible air leak, inflating the cuff with minimal occlusive pressure to a peak inflation pressure of 20-22 cmH2O during positive pressure ventilation, inflating the cuff until the airway is closed by maintaining a continuous positive airway pressure of 20 cmH2O, or cuff manometers are commonly used applications. Although cuff manometers can be used to guide the monitoring of cuff pressure, their use and availability is not mandatory in many institutions around the world (due to the large number of anaesthetic areas, it is not possible to have a manometer everywhere). Therefore, in anaesthetic practice, cuff pressure is monitored manually or using a manometer at regular intervals during the operation.

Aim/Hypothesis:

H0: Endotracheal tube cuff pressure does not change with hyperextension position given to the neck during adenoidectomy, tonsillectomy or adenotonsillectomy surgery.

H1: Endotracheal tube cuff pressure changes with hyperextension position given to the neck during adenoidectomy, tonsillectomy or adenotonsillectomy surgery.

Material-Methods: The study will include patients between the ages of 2-18 years who will undergo adenoidectomy, tonsillectomy or adenotonsillectomy after obtaining informed consent from their parents. Routine practice will be followed for induction and maintenance of anaesthesia. Patients monitored in the operating room according to the standard American Society of Anesthesiologists (ASA) protocol will be orotracheally intubated with an ETT of appropriate internal diameter after induction of anaesthesia by the anaesthesiologist responsible for the patient. After the tube placement of the intubated patients is confirmed by the responsible anaesthesiologist, the ETT cuff will be measured and recorded by the responsible investigator with a cuff manometer (VBM Medizintechnik, GmbH, Germany) while the head and neck are in the neutral position (T0). When the patients are given the head-neck hyperextension position in which the surgery will be performed by the surgical team responsible for the patient's surgery, the pressure measurements will be repeated by the responsible investigator (T1). At the end of the operation, when the head and neck are returned to the neutral position, the tubular cuff pressure will be measured by the responsible investigator for the last time (T2).

Patients between 2-18 years of age who underwent adenoidectomy, tonsillectomy or adenotonsillectomy surgery will be included in the study. Patients with head and neck mobility restriction, patients who have had neck surgery before, and patients with body mass index (BMI) > 35 kg/m2 will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2-18 years
* undergoing adenoidectomy, tonsillectomy or adenotonsillectomy surgery

Exclusion Criteria:

* Patients with restricted head and neck mobility,
* patients with intraoperative complications,
* patients with previous neck surgery,
* patients with BMI > 35 kg/m2

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sample size was calculated using G*Power software, version 3.1.9.6. The effect size used in the calculation was derived from the study conducted by Kako et al. in which head position and cuff pressure changes were compared in the paediatric age group. Kako et al. reported that the cuff pressure was 18.3 ± 6.6 cmH2O in the neutral position and 20.9 ± 10.5 cmH2O when the head was extended (effect size 0.23). According to these data, a minimum sample size of 120 patients with a type-1 error level of 0.05, an effect size of 0.23 and a working power of 80% was calculated to determine the difference in cuff pressure with head position.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cuff pressure | intraoperative 3 times
  Intubation tube cuff pressure in cmH2O at 3 different time periods with a cuff manometer (VBM Medizintechnik, GmbH, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Erbil Türksal, Specialist, Principal Investigator — University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital
Locations (1):
- University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No